CLINICAL TRIAL: NCT05022784
Title: Real-World Medication Adherence Trajectories to Nintedanib Among Idiopathic Pulmonary Fibrosis Patients
Brief Title: Adherence to Nintedanib Among Idiopathic Pulmonary Fibrosis Patients
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1199-0471
Record Dates: First submitted 2021-08-20; First posted 2021-08-26 (Actual); Results first posted 2024-04-19 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2023-11

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — nintedanib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Idiopathic Pulmonary Fibrosis Patients: Medicare beneficiaries with IPF who newly initiated treatment with nintedanib
  Interventions: Drug: Nintedanib

INTERVENTIONS:
Drug: Nintedanib — Nintedanib

SUMMARY:
This is a non-interventional cohort study using existing administrative data from the U.S. Medicare program.

This study has two objectives:

* Identification of adherence trajectories of nintedanib among Idiopathic Pulmonary Fibrosis (IPF) patients.
* Understanding characteristics of patients within each nintedanib adherence trajectory among IPF patients.

ELIGIBILITY:
Inclusion criteria:

* Newly initiated nintedanib during 10/01/2014 to 12/31/2018
* Were at least 66 years old as of the date of their first nintedanib prescription claim (index date)
* Qualified for Medicare based on age
* Had at least 12 months (365 days) of continuous enrollment in Medicare Parts A, B and D before (baseline period) and 12 months (360 days) after the index date (follow-up period)
* Had at least one inpatient or two outpatient claims (>14 days apart) with a diagnosis code for Idiopathic Pulmonary Fibrosis (IPF) during the baseline period

Exclusion criteria:

* Had any history of pirfenidone or nintedanib use during the baseline period
* Had any history of lung transplant during the baseline, index date or follow-up periods
* Had any claims for skilled nursing facility, long-term care facility or hospice during the baseline, index date or follow-up period
* Had evidence during the baseline period of any of the following conditions: lung cancer, autoimmune, or connective tissue diseases (i.e. rheumatoid arthritis (RA), sarcoidosis, systemic lupus erythematosus (SLE), dermatopolymyositis, systemic sclerosis, Sjogren's, and mixed connective tissue disease (CTD)) during the baseline period
* Had dual eligibility of Medicare and Medicaid
* Had history of using pirfenidone at the same time with nintedanib during follow-up

Min Age: 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The study sample will consist of community-dwelling Medicare beneficiaries with Idiopathic Pulmonary Fibrosis (IPF) who initiate treatment with nintedanib.
Sampling Method: Non-Probability Sample
Enrollment: 1798 (Actual)
Dates: Start 2021-08-23 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Medicus Economics, LCC, Milton, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A Real world, non-interventional study based on existing data from administrative enrollment and claims data from the United States (U.S.) federal Medicare program for beneficiaries who were continuously enrolled in Original Medicare insurance coverage. The study aimed to identify adherence trajectories of nintedanib use among Idiopathic Pulmonary Fibrosis (IPF) patients and to understand characteristics of patients within each nintedanib adherence trajectory among IPF patients.
Pre-assignment Details: Only subjects that met all inclusion and none of the exclusion criteria were included.
Groups:
- Nintedanib: This arm included Idiopathic Pulmonary Fibrosis (IPF) patients who newly initiated treatment with nintedanib between 1st October 2014 and 31st December 2018.
Period: Overall Study
Arm/Group | Nintedanib
Started | 1798
Eligible Patients | 1798
Completed | 1798
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Eligible Patients set: All patients who met the criteria were included in the analysis dataset.
Arm/Group | Nintedanib
Number analyzed (Participants) | 1798
Age, Continuous [Mean (Standard Deviation); unit: Years] | 75.40 (5.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 700
  Male | 1098
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian/Pacific Isla | 29
  Black | 36
  Hispanic | 61
  Non-Hispanic White | 1638
  Other/Missing | 34

OUTCOME MEASURES:

1. Primary Outcome: Adherence Trajectories to Nintedanib Among Idiopathic Pulmonary Fibrosis (IPF) Patients
Description: The number of IPF patients per adherence trajectories to nintedanib is presented. The first claim for nintedanib was used for defining the initiation date. For each 30-day month (12 months) following the nintedanib initiation date, the Proportions of Days Covered (PDC) were calculated as the sum of days with supply divided by 30, the monthly nintedanib proportion of days covered was then calculated. The twelve 30-days PDC values were used as outcomes in the Group-based trajectory model (GBTM), the probabilities that a given individual is in each of the latent clusters was calculated by the GBTM estimation procedure using the monthly binary PDC ≥ 0.8 indicators as outcomes.
  The reported types of trajectories to nintedanib were:
  * Highly adherent (PDC ≈ 0.9)
  * Medium adherent (PDC ≈ 0.4-0.6) - Gradual decliners (PDC bottoms out by month 11)
  * Intermediate decliners (PDC bottoms out by month 8)
  * Rapid decliners (PDC approaches zero by month 4)
Time Frame: Up to 1 year
Population: Eligible Patients set: All patients who met the criteria were included in the analysis dataset.
Measure: Count of Participants; unit: Participants
Arm/Group | Nintedanib
Number analyzed (Participants) | 1798
Participants
  Highly adherent | 781
  Medium adherent | 202
  Gradual decliners | 190
  Intermediate decliners | 255
  Rapid decliners | 370

2. Secondary Outcome: Demographic Characteristic: Age According to Adherence Trajectories for the Idiopathic Pulmonary Fibrosis (IPF) Patients Who Were Initiated on Nintedanib
Description: Age according to adherence trajectories for the idiopathic pulmonary fibrosis (IPF) patients who were initiated on nintedanib is reported. Age for each patient was calculated by subtracting the year of birth from the year of index (i.e. Year of the index date- Year of birth). Year of index was defined as the year the patients where initiated on nintedanib treatment.
Time Frame: Baseline period: 360 consecutive days ending the day before the index date (i.e., the date of the patient's first claim for nintedanib). Up to 360 days.
Population: Eligible Patients set: All patients who met the criteria were included in the analysis dataset.
Measure: Mean (Standard Deviation); unit: Years
Groups:
- Nintedanib- Highly Adherent: This trajectory included highly adherent Idiopathic Pulmonary Fibrosis (IPF) patients who newly initiated treatment with nintedanib between 1st October 2014 and 31st December 2018. Proportions of Days Covered (PDC) ≈ 0.9.
- Nintedanib- Medium Adherent: This trajectory included Medium adherent Idiopathic Pulmonary Fibrosis (IPF) patients who newly initiated treatment with nintedanib between 1st October 2014 and 31st December 2018. Proportions of Days Covered (PDC ≈ 0.4-0.6).
- Nintedanib- Gradual Decliners: This trajectory included Gradual decliners Idiopathic Pulmonary Fibrosis (IPF) patients who newly initiated treatment with nintedanib between 1st October 2014 and 31st December 2018. Proportions of Days Covered (PDC bottoms out by month 11).
- Nintedanib- Intermediate Decliners: This trajectory included Intermediate decliners Idiopathic Pulmonary Fibrosis (IPF) patients who newly initiated treatment with nintedanib between 1st October 2014 and 31st December 2018. Proportions of Days Covered (PDC bottoms out by month 8).
- Nintedanib- Rapid Decliners: This trajectory included Rapid decliners Idiopathic Pulmonary Fibrosis (IPF) patients who newly initiated treatment with nintedanib between 1st October 2014 and 31st December 2018. Proportions of Days Covered (PDC approaches zero by month 4).
Arm/Group | Nintedanib- Highly Adherent | Nintedanib- Medium Adherent | Nintedanib- Gradual Decliners | Nintedanib- Intermediate Decliners | Nintedanib- Rapid Decliners
Number analyzed (Participants) | 781 | 202 | 190 | 255 | 370
Years | 74.65 (5.36) | 75.21 (5.45) | 75.89 (5.60) | 76.29 (5.61) | 76.21 (5.62)
Statistical Analysis 1: Comparison: Nintedanib- Highly Adherent vs Nintedanib- Medium Adherent vs Nintedanib- Gradual Decliners vs Nintedanib- Intermediate Decliners vs Nintedanib- Rapid Decliners; The statistical method applied in this analysis is Analysis of Variance (ANOVA), which compares the mean value in each group and tests if they are significantly different via a fixed-effect regression model; Test type: Other; p < .0001, ANOVA

3. Secondary Outcome: Demographic Characteristic: Sex According to Adherence Trajectories for the Idiopathic Pulmonary Fibrosis (IPF) Patients Who Were Initiated on Nintedanib
Description: Number of patients per sex according to adherence trajectories for the idiopathic pulmonary fibrosis (IPF) patients who were initiated on nintedanib is reported.
Time Frame: Data collected at the study index date, i.e., the date of the patient's first claim for nintedanib.
Population: Eligible Patients set: All patients who met the criteria were included in the analysis dataset.
Measure: Count of Participants; unit: Participants
Arm/Group | Nintedanib- Highly Adherent | Nintedanib- Medium Adherent | Nintedanib- Gradual Decliners | Nintedanib- Intermediate Decliners | Nintedanib- Rapid Decliners
Number analyzed (Participants) | 781 | 202 | 190 | 255 | 370
Participants
  Male | 530 | 113 | 124 | 138 | 193
  Female | 251 | 89 | 66 | 117 | 177
Statistical Analysis 1: Comparison: Nintedanib- Highly Adherent vs Nintedanib- Medium Adherent vs Nintedanib- Gradual Decliners vs Nintedanib- Intermediate Decliners vs Nintedanib- Rapid Decliners; The statistical method applied in this analysis is Chi-squared hypothesis test, which tested if the count in each group was impacted by any confounding variable; Test type: Other; p < .0001, Chi-squared

4. Secondary Outcome: Demographic Characteristic: Race/Ethnicity According to Adherence Trajectories for the Idiopathic Pulmonary Fibrosis (IPF) Patients Who Were Initiated on Nintedanib
Description: Number of patients per Race/ethnicity according to adherence trajectories for the idiopathic pulmonary fibrosis (IPF) patients who were initiated on nintedanib is reported.
Time Frame: Data collected at the study index date, i.e., the date of the patient's first claim for nintedanib.
Population: Eligible Patients set: All patients who met the criteria were included in the analysis dataset.
Measure: Count of Participants; unit: Participants
Arm/Group | Nintedanib- Highly Adherent | Nintedanib- Medium Adherent | Nintedanib- Gradual Decliners | Nintedanib- Intermediate Decliners | Nintedanib- Rapid Decliners
Number analyzed (Participants) | 781 | 202 | 190 | 255 | 370
Participants
  White non-Hispanic | 718 | 183 | 171 | 237 | 329
  Non-White | 63 | 19 | 19 | 18 | 41
Statistical Analysis 1: Comparison: Nintedanib- Highly Adherent vs Nintedanib- Medium Adherent vs Nintedanib- Gradual Decliners vs Nintedanib- Intermediate Decliners vs Nintedanib- Rapid Decliners; [analysis description as in outcome 3, analysis 1]; Test type: Other; p = 0.37, Chi-squared

5. Secondary Outcome: Demographic Characteristic: Census Region According to Adherence Trajectories for the Idiopathic Pulmonary Fibrosis (IPF) Patients Who Were Initiated on Nintedanib
Description: Number of patients per census region according to adherence trajectories for the idiopathic pulmonary fibrosis (IPF) patients who were initiated on nintedanib is reported. The beneficiary's state of residence into Census regions (Northeast, South, Midwest, West and Puerto Rico) from the enrollment record and covering the index date.
Time Frame: Data collected at the study index date, i.e., the date of the patient's first claim for nintedanib.
Population: Eligible Patients set: All patients who met the criteria were included in the analysis dataset.
Measure: Count of Participants; unit: Participants
Arm/Group | Nintedanib- Highly Adherent | Nintedanib- Medium Adherent | Nintedanib- Gradual Decliners | Nintedanib- Intermediate Decliners | Nintedanib- Rapid Decliners
Number analyzed (Participants) | 781 | 202 | 190 | 255 | 370
Participants
  Midwest | 172 | 46 | 51 | 55 | 92
  Northeast | 104 | 31 | 27 | 48 | 46
  South and Puerto Rico | 344 | 84 | 79 | 113 | 171
  West | 161 | 41 | 33 | 39 | 61
Statistical Analysis 1: Comparison: Nintedanib- Highly Adherent vs Nintedanib- Medium Adherent vs Nintedanib- Gradual Decliners vs Nintedanib- Intermediate Decliners vs Nintedanib- Rapid Decliners; [analysis description as in outcome 3, analysis 1]; Test type: Other; p = 0.477, Chi-squared

6. Secondary Outcome: Demographic Characteristic: Social Deprivation Index According to Adherence Trajectories for the Idiopathic Pulmonary Fibrosis (IPF) Patients Who Were Initiated on Nintedanib
Description: Social deprivation index according to adherence trajectories for the idiopathic pulmonary fibrosis (IPF) patients who were initiated on nintedanib is reported. Social deprivation index (SDI) was a continuous variable and ranged between 0 and 100 representing the SDI for the beneficiary's residential ZIP Code. Higher values for the SDI indicate more social deprivation. The SDI was calculated as a composite measure of seven demographic characteristics collected in the American Community Survey (ACS): percent living in poverty, percent with less than 12 years of education, percent single parent household, percent living in rented housing unit, percent living in overcrowded housing unit, percent of households without a car, and percent non-employed adults under 65 years of age.
Time Frame: Data collected at the study index date, i.e., the date of the patient's first claim for nintedanib.
Population: Eligible Patients set: All patients who met the criteria were included in the analysis dataset.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Nintedanib- Highly Adherent | Nintedanib- Medium Adherent | Nintedanib- Gradual Decliners | Nintedanib- Intermediate Decliners | Nintedanib- Rapid Decliners
Number analyzed (Participants) | 781 | 202 | 190 | 255 | 370
Units on a scale | 41.63 (25.65) | 39.27 (25.10) | 39.61 (26.01) | 39.61 (25.81) | 40.20 (25.77)
Statistical Analysis 1: Comparison: Nintedanib- Highly Adherent vs Nintedanib- Medium Adherent vs Nintedanib- Gradual Decliners vs Nintedanib- Intermediate Decliners vs Nintedanib- Rapid Decliners; The statistical method applied in this analysis is Analysis of Variance (ANOVA), which compared the mean value in each group and tests if they are significantly different via a fixed-effect regression model; Test type: Other; p = 0.644, ANOVA

7. Secondary Outcome: Clinical Characteristic: Combined Comorbidity Index According to Adherence Trajectories for the Idiopathic Pulmonary Fibrosis (IPF) Patients Who Were Initiated on Nintedanib
Description: Combined comorbidity index (CCI) according to adherence trajectories for the idiopathic pulmonary fibrosis (IPF) patients who were initiated on nintedanib is reported. The CCI Gagne et al.'s (2011) scored ranging from 0 to 26 measured from comorbidity diagnosis codes on inpatient, outpatient and Carrier claims that occurred during the baseline period, Higher scores indicated a more severe condition. The 20 conditions (with their weights in parentheses) include: Metastatic cancer (5), Congestive heart failure (2), Dementia (2), Renal failure (2), Weight loss (2), Hemiplegia (1), Alcohol abuse (1), Any tumor (1), Cardiac arrhythmias (1), Chronic pulmonary disease (1), Coagulopathy (1), Complicated diabetes (1), Deficiency anemia (1), Fluid and electrolyte disorders (1), Liver disease (1), Peripheral vascular disease (1), Psychosis (1), Pulmonary circulation disorders (1), HIV/AIDS (-1), and Hypertension (-1). The cumulative weight of the 20 conditions yields the CCI.
Time Frame: as for outcome 2
Population: Eligible Patients set: All patients who met the criteria were included in the analysis dataset.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nintedanib- Highly Adherent | Nintedanib- Medium Adherent | Nintedanib- Gradual Decliners | Nintedanib- Intermediate Decliners | Nintedanib- Rapid Decliners
Number analyzed (Participants) | 781 | 202 | 190 | 255 | 370
score on a scale | 2.86 (2.58) | 2.91 (2.54) | 2.85 (2.37) | 3.14 (2.46) | 3.19 (2.59)
Statistical Analysis 1: Comparison: Nintedanib- Highly Adherent vs Nintedanib- Medium Adherent vs Nintedanib- Gradual Decliners vs Nintedanib- Intermediate Decliners vs Nintedanib- Rapid Decliners; [analysis description as in outcome 6, analysis 1]; Test type: Other; p = 0.206, ANOVA

8. Secondary Outcome: Clinical Characteristic: Combined Comorbidity Index According to Adherence Trajectories for the Idiopathic Pulmonary Fibrosis (IPF) Patients Who Were Initiated on Nintedanib
Description: Number of patients per Combined comorbidity index (CCI) according to adherence trajectories for the idiopathic pulmonary fibrosis (IPF) patients who were initiated on nintedanib is reported. The CCI Gagne et al.'s (2011) scored ranging from 0 to 26 as measured from comorbidity diagnosis codes in any position on inpatient, outpatient and Carrier claims that occurred during the baseline period, higher scores indicated a more severe condition. The 20 conditions in the CCI (with their weights in parentheses) include: Metastatic cancer (5), Congestive heart failure (2), Dementia (2), Renal failure (2), Weight loss (2), Hemiplegia (1), Alcohol abuse (1), Any tumor (1), Cardiac arrhythmias (1), Chronic pulmonary disease (1), Coagulopathy (1), Complicated diabetes (1), Deficiency anemia (1), Fluid and electrolyte disorders (1), Liver disease (1), Peripheral vascular disease (1), Psychosis (1), Pulmonary circulation disorders (1), HIV/AIDS (-1), and Hypertension (-1).
Time Frame: as for outcome 2
Population: Eligible Patients set: All patients who met the criteria were included in the analysis dataset.
Measure: Number; unit: score on a scale
Arm/Group | Nintedanib- Highly Adherent | Nintedanib- Medium Adherent | Nintedanib- Gradual Decliners | Nintedanib- Intermediate Decliners | Nintedanib- Rapid Decliners
Number analyzed (Participants) | 781 | 202 | 190 | 255 | 370
score on a scale
  0 | 139 | 45 | 32 | 33 | 55
  1 | 156 | 25 | 37 | 37 | 62
  2 | 118 | 32 | 29 | 43 | 55
  3 | 117 | 30 | 22 | 52 | 49
  4 | 73 | 19 | 28 | 30 | 45
  5+ | 178 | 51 | 42 | 60 | 104
Statistical Analysis 1: Comparison: Nintedanib- Highly Adherent vs Nintedanib- Medium Adherent vs Nintedanib- Gradual Decliners vs Nintedanib- Intermediate Decliners vs Nintedanib- Rapid Decliners; [analysis description as in outcome 3, analysis 1]; Test type: Other; p = 0.052, Chi-squared

9. Secondary Outcome: Clinical Characteristic: Congestive Heart Failure According to Adherence Trajectories for the Idiopathic Pulmonary Fibrosis (IPF) Patients Who Were Initiated on Nintedanib
Description: Number of patients with diagnosis of Congestive heart failure according to adherence trajectories for the idiopathic pulmonary fibrosis (IPF) patients who were initiated on nintedanib is reported. A binary indicator for whether the beneficiary had a diagnosis code for Congestive heart failure on at least one inpatient, outpatient or Carrier claim that occurred during the baseline period.
Time Frame: as for outcome 2
Population: Eligible Patients set: All patients who met the criteria were included in the analysis dataset.
Measure: Count of Participants; unit: Participants
Arm/Group | Nintedanib- Highly Adherent | Nintedanib- Medium Adherent | Nintedanib- Gradual Decliners | Nintedanib- Intermediate Decliners | Nintedanib- Rapid Decliners
Number analyzed (Participants) | 781 | 202 | 190 | 255 | 370
Participants
  Yes | 257 | 65 | 53 | 101 | 140
  No | 524 | 137 | 137 | 154 | 230
Statistical Analysis 1: Comparison: Nintedanib- Highly Adherent vs Nintedanib- Medium Adherent vs Nintedanib- Gradual Decliners vs Nintedanib- Intermediate Decliners vs Nintedanib- Rapid Decliners; [analysis description as in outcome 3, analysis 1]; Test type: Other; p = 0.044, Chi-squared

10. Secondary Outcome: Clinical Characteristic: Renal Failure According to Adherence Trajectories for the Idiopathic Pulmonary Fibrosis (IPF) Patients Who Were Initiated on Nintedanib
Description: Number of patients with diagnosis of Renal failure according to adherence trajectories for the idiopathic pulmonary fibrosis (IPF) patients who were initiated on nintedanib is reported. A binary indicator for whether the beneficiary had a diagnosis code for Renal failure on at least one inpatient, outpatient or Carrier claim that occurred during the baseline period.
Time Frame: Data collected at Baseline period: 360 consecutive days ending the day before the index date (i.e., the date of the patient's first claim for nintedanib). Up to 360 days.
Population: Eligible Patients set: All patients who met the criteria were included in the analysis dataset.
Measure: Count of Participants; unit: Participants
Arm/Group | Nintedanib- Highly Adherent | Nintedanib- Medium Adherent | Nintedanib- Gradual Decliners | Nintedanib- Intermediate Decliners | Nintedanib- Rapid Decliners
Number analyzed (Participants) | 781 | 202 | 190 | 255 | 370
Participants
  Diagnosed Renal failure | 116 | 40 | 31 | 39 | 62
  Not Diagnosed Renal failure | 665 | 162 | 159 | 216 | 308
Statistical Analysis 1: Comparison: Nintedanib- Highly Adherent vs Nintedanib- Medium Adherent vs Nintedanib- Gradual Decliners vs Nintedanib- Intermediate Decliners vs Nintedanib- Rapid Decliners; [analysis description as in outcome 3, analysis 1]; Test type: Other; p = 0.525, Chi-squared

11. Secondary Outcome: Clinical Characteristic: Cardiac Arrhythmias According to Adherence Trajectories for the Idiopathic Pulmonary Fibrosis (IPF) Patients Who Were Initiated on Nintedanib
Description: Number of patients with diagnosis of Cardiac arrhythmias according to adherence trajectories for the idiopathic pulmonary fibrosis (IPF) patients who were initiated on nintedanib is reported. A binary indicator for whether the beneficiary had a diagnosis code for Cardiac arrhythmias on at least one inpatient, outpatient or Carrier claim that occurred during the baseline period.
Time Frame: as for outcome 2
Population: Eligible Patients set: All patients who met the criteria were included in the analysis dataset.
Measure: Count of Participants; unit: Participants
Arm/Group | Nintedanib- Highly Adherent | Nintedanib- Medium Adherent | Nintedanib- Gradual Decliners | Nintedanib- Intermediate Decliners | Nintedanib- Rapid Decliners
Number analyzed (Participants) | 781 | 202 | 190 | 255 | 370
Participants
  Diagnosed cardiac arrhythmias | 232 | 60 | 72 | 84 | 141
  Not diagnosed Cardiac arrhythmias | 549 | 142 | 118 | 171 | 229
Statistical Analysis 1: Comparison: Nintedanib- Highly Adherent vs Nintedanib- Medium Adherent vs Nintedanib- Gradual Decliners vs Nintedanib- Intermediate Decliners vs Nintedanib- Rapid Decliners; [analysis description as in outcome 3, analysis 1]; Test type: Other; p = 0.024, Chi-squared

12. Secondary Outcome: Clinical Characteristic: Peripheral Vascular Disease According to Adherence Trajectories for the Idiopathic Pulmonary Fibrosis (IPF) Patients Who Were Initiated on Nintedanib
Description: Number of patients with diagnosis of Peripheral vascular disease according to adherence trajectories for the idiopathic pulmonary fibrosis (IPF) patients who were initiated on nintedanib is reported. A binary indicator for whether the beneficiary had a diagnosis code for Peripheral vascular disease on at least one inpatient, outpatient or Carrier claim that occurred during the baseline period.
Time Frame: as for outcome 2
Population: Eligible Patients set: All patients who met the criteria were included in the analysis dataset.
Measure: Count of Participants; unit: Participants
Arm/Group | Nintedanib- Highly Adherent | Nintedanib- Medium Adherent | Nintedanib- Gradual Decliners | Nintedanib- Intermediate Decliners | Nintedanib- Rapid Decliners
Number analyzed (Participants) | 781 | 202 | 190 | 255 | 370
Participants
  Peripheral vascular disease | 170 | 54 | 44 | 73 | 112
  No Peripheral vascular disease | 611 | 148 | 146 | 182 | 258
Statistical Analysis 1: Comparison: Nintedanib- Highly Adherent vs Nintedanib- Medium Adherent vs Nintedanib- Gradual Decliners vs Nintedanib- Intermediate Decliners vs Nintedanib- Rapid Decliners; [analysis description as in outcome 3, analysis 1]; Test type: Other; p = 0.016, Chi-squared

13. Secondary Outcome: Clinical Characteristic: Hypertension According to Adherence Trajectories for the Idiopathic Pulmonary Fibrosis (IPF) Patients Who Were Initiated on Nintedanib
Description: Number of patients with diagnosis of Hypertension according to adherence trajectories for the idiopathic pulmonary fibrosis (IPF) patients who were initiated on nintedanib is reported. A binary indicator for whether the beneficiary had a diagnosis code for Hypertension on at least one inpatient, outpatient or Carrier claim that occurred during the baseline period.
Time Frame: as for outcome 2
Population: Eligible Patients set: All patients who met the criteria were included in the analysis dataset.
Measure: Count of Participants; unit: Participants
Arm/Group | Nintedanib- Highly Adherent | Nintedanib- Medium Adherent | Nintedanib- Gradual Decliners | Nintedanib- Intermediate Decliners | Nintedanib- Rapid Decliners
Number analyzed (Participants) | 781 | 202 | 190 | 255 | 370
Participants
  Hypertension | 614 | 161 | 149 | 198 | 298
  No Hypertension | 167 | 41 | 41 | 57 | 72
Statistical Analysis 1: Comparison: Nintedanib- Highly Adherent vs Nintedanib- Medium Adherent vs Nintedanib- Gradual Decliners vs Nintedanib- Intermediate Decliners vs Nintedanib- Rapid Decliners; [analysis description as in outcome 3, analysis 1]; Test type: Other; p = 0.913, Chi-squared

14. Secondary Outcome: Clinical Characteristic- IPF Comorbid Conditions: Asthma According to Adherence Trajectories for the Idiopathic Pulmonary Fibrosis (IPF) Patients Who Were Initiated on Nintedanib
Description: Number of patients with diagnosis of Asthma according to adherence trajectories for the idiopathic pulmonary fibrosis (IPF) patients who were initiated on nintedanib is reported. A binary indicator for whether the beneficiary had a diagnosis code for Asthma on at least one inpatient, outpatient or Carrier claim that occurred during the baseline period.
Time Frame: as for outcome 2
Population: Eligible Patients set: All patients who met the criteria were included in the analysis dataset.
Measure: Count of Participants; unit: Participants
Arm/Group | Nintedanib- Highly Adherent | Nintedanib- Medium Adherent | Nintedanib- Gradual Decliners | Nintedanib- Intermediate Decliners | Nintedanib- Rapid Decliners
Number analyzed (Participants) | 781 | 202 | 190 | 255 | 370
Participants
  Asthma | 132 | 34 | 31 | 32 | 67
  No Asthma | 649 | 168 | 159 | 223 | 303
Statistical Analysis 1: Comparison: Nintedanib- Highly Adherent vs Nintedanib- Medium Adherent vs Nintedanib- Gradual Decliners vs Nintedanib- Intermediate Decliners vs Nintedanib- Rapid Decliners; [analysis description as in outcome 3, analysis 1]; Test type: Other; p = 0.448, Chi-squared

15. Secondary Outcome: Clinical Characteristic- IPF Comorbid Conditions: Chronic Obstructive Pulmonary Disease According to Adherence Trajectories for the Idiopathic Pulmonary Fibrosis (IPF) Patients Who Were Initiated on Nintedanib
Description: Number of patients with diagnosis of Chronic obstructive pulmonary disease according to adherence trajectories for the idiopathic pulmonary fibrosis (IPF) patients who were initiated on nintedanib is reported. A binary indicator for whether the beneficiary had a diagnosis code for Chronic obstructive pulmonary disease on at least one inpatient, outpatient or Carrier claim that occurred during the baseline period.
Time Frame: as for outcome 2
Population: Eligible Patients set: All patients who met the criteria were included in the analysis dataset.
Measure: Count of Participants; unit: Participants
Groups:
- Nintedanib- Rapid Decliners: Nintedanib- Rapid decliners 370 This trajectory included Rapid decliners Idiopathic Pulmonary Fibrosis (IPF) patients who newly initiated treatment with nintedanib between 1st October 2014 and 31st December 2018. Proportions of Days Covered (PDC approaches zero by month 4).
Arm/Group | Nintedanib- Highly Adherent | Nintedanib- Medium Adherent | Nintedanib- Gradual Decliners | Nintedanib- Intermediate Decliners | Nintedanib- Rapid Decliners
Number analyzed (Participants) | 781 | 202 | 190 | 255 | 370
Participants
  Chronic obstructive pulmonary disease | 373 | 86 | 86 | 115 | 183
  No Chronic obstructive pulmonary disease | 408 | 116 | 104 | 140 | 187
Statistical Analysis 1: Comparison: Nintedanib- Highly Adherent vs Nintedanib- Medium Adherent vs Nintedanib- Gradual Decliners vs Nintedanib- Intermediate Decliners vs Nintedanib- Rapid Decliners; [analysis description as in outcome 3, analysis 1]; Test type: Other; p = 0.515, Chi-squared

16. Secondary Outcome: Clinical Characteristic- IPF Comorbid Conditions: Gastroesophageal Reflux Disease According to Adherence Trajectories for the Idiopathic Pulmonary Fibrosis (IPF) Patients Who Were Initiated on Nintedanib
Description: Number of patients with diagnosis of Gastroesophageal reflux disease according to adherence trajectories for the idiopathic pulmonary fibrosis (IPF) patients who were initiated on nintedanib is reported. A binary indicator for whether the beneficiary had a diagnosis code for Gastroesophageal reflux disease on at least one inpatient, outpatient or Carrier claim that occurred during the baseline period.
Time Frame: as for outcome 2
Population: Eligible Patients set: All patients who met the criteria were included in the analysis dataset.
Measure: Count of Participants; unit: Participants
Groups:
- Nintedanib- Gradual Decliners: Nintedanib- Gradual decliners 190 This trajectory included Gradual decliners Idiopathic Pulmonary Fibrosis (IPF) patients who newly initiated treatment with nintedanib between 1st October 2014 and 31st December 2018. Proportions of Days Covered (PDC bottoms out by month 11).
Arm/Group | Nintedanib- Highly Adherent | Nintedanib- Medium Adherent | Nintedanib- Gradual Decliners | Nintedanib- Intermediate Decliners | Nintedanib- Rapid Decliners
Number analyzed (Participants) | 781 | 202 | 190 | 255 | 370
Participants
  Gastroesophageal reflux disease | 398 | 104 | 97 | 125 | 199
  No Gastroesophageal reflux disease | 383 | 98 | 93 | 130 | 171
Statistical Analysis 1: Comparison: Nintedanib- Highly Adherent vs Nintedanib- Medium Adherent vs Nintedanib- Gradual Decliners vs Nintedanib- Intermediate Decliners vs Nintedanib- Rapid Decliners; [analysis description as in outcome 3, analysis 1]; Test type: Other; p = 0.829, Chi-squared

17. Secondary Outcome: Clinical Characteristic- IPF Comorbid Conditions: Hypoxia According to Adherence Trajectories for the Idiopathic Pulmonary Fibrosis (IPF) Patients Who Were Initiated on Nintedanib
Description: Number of patients with diagnosis of Hypoxia according to adherence trajectories for the idiopathic pulmonary fibrosis (IPF) patients who were initiated on nintedanib is reported. A binary indicator for whether the beneficiary had a diagnosis code for Hypoxia on at least one inpatient, outpatient or Carrier claim that occurred during the baseline period.
Time Frame: as for outcome 2
Population: Eligible Patients set: All patients who met the criteria were included in the analysis dataset.
Measure: Count of Participants; unit: Participants
Arm/Group | Nintedanib- Highly Adherent | Nintedanib- Medium Adherent | Nintedanib- Gradual Decliners | Nintedanib- Intermediate Decliners | Nintedanib- Rapid Decliners
Number analyzed (Participants) | 781 | 202 | 190 | 255 | 370
Participants
  Hypoxia | 234 | 57 | 63 | 83 | 100
  No Hypoxia | 547 | 145 | 127 | 172 | 270
Statistical Analysis 1: Comparison: Nintedanib- Highly Adherent vs Nintedanib- Medium Adherent vs Nintedanib- Gradual Decliners vs Nintedanib- Intermediate Decliners vs Nintedanib- Rapid Decliners; [analysis description as in outcome 3, analysis 1]; Test type: Other; p = 0.471, Chi-squared

18. Secondary Outcome: Clinical Characteristic- IPF Comorbid Conditions: Pulmonary Hypertension According to Adherence Trajectories for the Idiopathic Pulmonary Fibrosis (IPF) Patients Who Were Initiated on Nintedanib
Description: Number of patients with diagnosis of Pulmonary hypertension according to adherence trajectories for the idiopathic pulmonary fibrosis (IPF) patients who were initiated on nintedanib is reported. A binary indicator for whether the beneficiary had a diagnosis code for Pulmonary hypertension on at least one inpatient, outpatient or Carrier claim that occurred during the baseline period.
Time Frame: as for outcome 2
Population: Eligible Patients set: All patients who met the criteria were included in the analysis dataset.
Measure: Count of Participants; unit: Participants
Arm/Group | Nintedanib- Highly Adherent | Nintedanib- Medium Adherent | Nintedanib- Gradual Decliners | Nintedanib- Intermediate Decliners | Nintedanib- Rapid Decliners
Number analyzed (Participants) | 781 | 202 | 190 | 255 | 370
Participants
  Pulmonary hypertension | 156 | 36 | 39 | 48 | 77
  No Pulmonary hypertension | 625 | 166 | 151 | 207 | 293
Statistical Analysis 1: Comparison: Nintedanib- Highly Adherent vs Nintedanib- Medium Adherent vs Nintedanib- Gradual Decliners vs Nintedanib- Intermediate Decliners vs Nintedanib- Rapid Decliners; [analysis description as in outcome 3, analysis 1]; Test type: Other; p = 0.915, Chi-squared

19. Secondary Outcome: Clinical Characteristic- IPF Comorbid Conditions: Sleep Apnea According to Adherence Trajectories for the Idiopathic Pulmonary Fibrosis (IPF) Patients Who Were Initiated on Nintedanib
Description: Number of patients with diagnosis of Sleep apnea according to adherence trajectories for the idiopathic pulmonary fibrosis (IPF) patients who were initiated on nintedanib is reported. A binary indicator for whether the beneficiary had a diagnosis code for Sleep apnea on at least one inpatient, outpatient or Carrier claim that occurred during the baseline period.
Time Frame: as for outcome 2
Population: Eligible Patients set: All patients who met the criteria were included in the analysis dataset.
Measure: Count of Participants; unit: Participants
Arm/Group | Nintedanib- Highly Adherent | Nintedanib- Medium Adherent | Nintedanib- Gradual Decliners | Nintedanib- Intermediate Decliners | Nintedanib- Rapid Decliners
Number analyzed (Participants) | 781 | 202 | 190 | 255 | 370
Participants
  Sleep apnea | 243 | 52 | 57 | 62 | 115
  No Sleep apnea | 538 | 150 | 133 | 193 | 255
Statistical Analysis 1: Comparison: Nintedanib- Highly Adherent vs Nintedanib- Medium Adherent vs Nintedanib- Gradual Decliners vs Nintedanib- Intermediate Decliners vs Nintedanib- Rapid Decliners; Test type: Other; p = 0.190, Chi-squared

20. Secondary Outcome: Clinical Characteristic- IPF Medical Services: High-res CT (High-resolution Computed Tomography) Scan According to Adherence Trajectories for the Idiopathic Pulmonary Fibrosis (IPF) Patients Who Were Initiated on Nintedanib
Description: Number of patients that used the medical service: High-res CT (High-resolution computed tomography) scan according to adherence trajectories for the idiopathic pulmonary fibrosis (IPF) patients who were initiated on nintedanib is reported. A binary indicator for whether the beneficiary had been performed a High-res CT scan on at least one inpatient, outpatient or Carrier claim that occurred during the baseline period.
Time Frame: as for outcome 2
Population: Eligible Patients set: All patients who met the criteria were included in the analysis dataset.
Measure: Count of Participants; unit: Participants
Arm/Group | Nintedanib- Highly Adherent | Nintedanib- Medium Adherent | Nintedanib- Gradual Decliners | Nintedanib- Intermediate Decliners | Nintedanib- Rapid Decliners
Number analyzed (Participants) | 781 | 202 | 190 | 255 | 370
Participants
  High-res CT scan | 597 | 157 | 144 | 200 | 280
  No High-res CT scan | 184 | 45 | 46 | 55 | 90
Statistical Analysis 1: Comparison: Nintedanib- Highly Adherent vs Nintedanib- Medium Adherent vs Nintedanib- Gradual Decliners vs Nintedanib- Intermediate Decliners vs Nintedanib- Rapid Decliners; [analysis description as in outcome 3, analysis 1]; Test type: Other; p = 0.928, Chi-squared

21. Secondary Outcome: Clinical Characteristic- IPF Medical Services: Lung Biopsy According to Adherence Trajectories for the Idiopathic Pulmonary Fibrosis (IPF) Patients Who Were Initiated on Nintedanib
Description: Number of patients that were performed a Lung biopsy according to adherence trajectories for the idiopathic pulmonary fibrosis (IPF) patients who were initiated on nintedanib is reported. A binary indicator for whether the beneficiary had a Lung biopsy biopsy on at least one inpatient, outpatient or Carrier claim that occurred during the baseline period.
Time Frame: as for outcome 2
Population: Eligible Patients set: All patients who met this criteria were included in the analysis dataset.
Measure: Count of Participants; unit: Participants
Arm/Group | Nintedanib- Highly Adherent | Nintedanib- Medium Adherent | Nintedanib- Gradual Decliners | Nintedanib- Intermediate Decliners | Nintedanib- Rapid Decliners
Number analyzed (Participants) | 781 | 202 | 190 | 255 | 370
Participants
  Lung biopsy | 134 | 37 | 26 | 35 | 64
  No Lung biopsy | 647 | 165 | 164 | 220 | 306
Statistical Analysis 1: Comparison: Nintedanib- Highly Adherent vs Nintedanib- Medium Adherent vs Nintedanib- Gradual Decliners vs Nintedanib- Intermediate Decliners vs Nintedanib- Rapid Decliners; [analysis description as in outcome 3, analysis 1]; Test type: Other; p = 0.490, Chi-squared

22. Secondary Outcome: Clinical Characteristic- IPF Medical Services: Oxygen Therapy or Supplemental Oxygen According to Adherence Trajectories for the Idiopathic Pulmonary Fibrosis (IPF) Patients Who Were Initiated on Nintedanib
Description: Number of patients that received Oxygen therapy or supplemental oxygen according to adherence trajectories for the idiopathic pulmonary fibrosis (IPF) patients who were initiated on nintedanib is reported. A binary indicator for whether the beneficiary received or not Oxygen therapy or supplemental oxygen on at least one inpatient, outpatient or Carrier claim that occurred during the baseline period.
Time Frame: as for outcome 2
Population: Eligible Patients set: All patients who met the criteria were included in the analysis dataset.
Measure: Count of Participants; unit: Participants
Arm/Group | Nintedanib- Highly Adherent | Nintedanib- Medium Adherent | Nintedanib- Gradual Decliners | Nintedanib- Intermediate Decliners | Nintedanib- Rapid Decliners
Number analyzed (Participants) | 781 | 202 | 190 | 255 | 370
Participants
  Oxygen therapy or supplemental oxygen | 128 | 28 | 32 | 45 | 69
  No Oxygen therapy or supplemental oxygen | 653 | 174 | 158 | 210 | 301
Statistical Analysis 1: Comparison: Nintedanib- Highly Adherent vs Nintedanib- Medium Adherent vs Nintedanib- Gradual Decliners vs Nintedanib- Intermediate Decliners vs Nintedanib- Rapid Decliners; [analysis description as in outcome 3, analysis 1]; Test type: Other; p = 0.667, Chi-squared

23. Secondary Outcome: Beneficiary Characteristics - Baseline HCRU (Health Care Resource Utilization) and Spending: Medication Count According to Adherence Trajectories for the Idiopathic Pulmonary Fibrosis (IPF) Patients Who Were Initiated on Nintedanib
Description: Medication count of the number of unique outpatient prescription medications for which beneficiary had claims during the baseline period, according to adherence trajectories for the idiopathic pulmonary fibrosis (IPF) patients who were initiated on nintedanib is reported.
Time Frame: as for outcome 2
Population: Eligible Patients set: All patients who met the criteria were included in the analysis dataset.
Measure: Mean (Standard Deviation); unit: Unique prescription medications
Arm/Group | Nintedanib- Highly Adherent | Nintedanib- Medium Adherent | Nintedanib- Gradual Decliners | Nintedanib- Intermediate Decliners | Nintedanib- Rapid Decliners
Number analyzed (Participants) | 781 | 202 | 190 | 255 | 370
Unique prescription medications | 10.94 (5.45) | 11.38 (5.87) | 11.57 (5.59) | 12.04 (5.69) | 11.77 (5.41)
Statistical Analysis 1: Comparison: Nintedanib- Highly Adherent vs Nintedanib- Medium Adherent vs Nintedanib- Gradual Decliners vs Nintedanib- Intermediate Decliners vs Nintedanib- Rapid Decliners; [analysis description as in outcome 6, analysis 1]; Test type: Other; p = 0.032, ANOVA

24. Secondary Outcome: Beneficiary Characteristics - Baseline HCRU (Health Care Resource Utilization) and Spending: Pharmacy Spending According to Adherence Trajectories for the Idiopathic Pulmonary Fibrosis (IPF) Patients Who Were Initiated on Nintedanib
Description: Total amount paid (Pharmacy spending) by all parties for outpatient prescription medications as reported in claims during the baseline period, according to adherence trajectories for the idiopathic pulmonary fibrosis (IPF) patients who were initiated on nintedanib is reported.
Time Frame: as for outcome 2
Population: Eligible Patients set: All patients who met the criteria were included in the analysis dataset.
Measure: Mean (Standard Deviation); unit: United States Dollar
Arm/Group | Nintedanib- Highly Adherent | Nintedanib- Medium Adherent | Nintedanib- Gradual Decliners | Nintedanib- Intermediate Decliners | Nintedanib- Rapid Decliners
Number analyzed (Participants) | 781 | 202 | 190 | 255 | 370
United States Dollar | 3,670 (10,951) | 3,042 (4,718) | 2,899 (4,078) | 3,711 (8,047) | 3,796 (9,229)
Statistical Analysis 1: Comparison: Nintedanib- Highly Adherent vs Nintedanib- Medium Adherent vs Nintedanib- Gradual Decliners vs Nintedanib- Intermediate Decliners vs Nintedanib- Rapid Decliners; [analysis description as in outcome 6, analysis 1]; Test type: Other; p = 0.721, ANOVA

25. Secondary Outcome: Beneficiary Characteristics - Baseline HCRU (Health Care Resource Utilization) and Spending: Pharmacy Spending - OOP According to Adherence Trajectories for the Idiopathic Pulmonary Fibrosis (IPF) Patients Who Were Initiated on Nintedanib
Description: The total amount paid out-of-pocket (Pharmacy spending - OOP) by the beneficiary for outpatient prescription medications as reported in Part D claims during the baseline period, according to adherence trajectories for the idiopathic pulmonary fibrosis (IPF) patients who were initiated on nintedanib is reported.
Time Frame: as for outcome 2
Population: Eligible Patients set: All patients who met the criteria were included in the analysis dataset.
Measure: Mean (Standard Error); unit: United States Dollar
Arm/Group | Nintedanib- Highly Adherent | Nintedanib- Medium Adherent | Nintedanib- Gradual Decliners | Nintedanib- Intermediate Decliners | Nintedanib- Rapid Decliners
Number analyzed (Participants) | 781 | 202 | 190 | 255 | 370
United States Dollar | 798 (1,062) | 732 (734) | 759 (801) | 807 (971) | 891 (1,019)
Statistical Analysis 1: Comparison: Nintedanib- Highly Adherent vs Nintedanib- Medium Adherent vs Nintedanib- Gradual Decliners vs Nintedanib- Intermediate Decliners vs Nintedanib- Rapid Decliners; [analysis description as in outcome 6, analysis 1]; Test type: Other; p = 0.352, ANOVA

26. Secondary Outcome: Beneficiary Characteristics - Inpatient Hospitalization Use and Spending: Inpatient Hospitalization According to Adherence Trajectories for the Idiopathic Pulmonary Fibrosis (IPF) Patients Who Were Initiated on Nintedanib
Description: Inpatient hospitalization was a binary indicator for whether a beneficiary had at least one inpatient hospitalization for any cause during the baseline period, according to adherence trajectories for the idiopathic pulmonary fibrosis (IPF) patients who were initiated on nintedanib is reported.
Time Frame: as for outcome 2
Population: Eligible Patients set: All patients who met the criteria were included in the analysis dataset.
Measure: Count of Participants; unit: Participants
Arm/Group | Nintedanib- Highly Adherent | Nintedanib- Medium Adherent | Nintedanib- Gradual Decliners | Nintedanib- Intermediate Decliners | Nintedanib- Rapid Decliners
Number analyzed (Participants) | 781 | 202 | 190 | 255 | 370
Participants
  No | 512 | 141 | 130 | 184 | 234
  Yes | 269 | 61 | 60 | 71 | 136
Statistical Analysis 1: Comparison: Nintedanib- Highly Adherent vs Nintedanib- Medium Adherent vs Nintedanib- Gradual Decliners vs Nintedanib- Intermediate Decliners vs Nintedanib- Rapid Decliners; [analysis description as in outcome 3, analysis 1]; Test type: Other; p = 0.136, Chi-squared

27. Secondary Outcome: Beneficiary Characteristics - Inpatient Hospitalization Use and Spending: Inpatient Hosp - Count According to Adherence Trajectories for the Idiopathic Pulmonary Fibrosis (IPF) Patients Who Were Initiated on Nintedanib
Description: The count of the number of inpatient hospitalizations for any cause a beneficiary had during the baseline period, according to adherence trajectories for the idiopathic pulmonary fibrosis (IPF) patients who were initiated on nintedanib is reported.
Time Frame: as for outcome 2
Population: Eligible Patients set: All patients who met the criteria were included in the analysis dataset.
Measure: Mean (Standard Deviation); unit: inpatient hospitalization
Arm/Group | Nintedanib- Highly Adherent | Nintedanib- Medium Adherent | Nintedanib- Gradual Decliners | Nintedanib- Intermediate Decliners | Nintedanib- Rapid Decliners
Number analyzed (Participants) | 781 | 202 | 190 | 255 | 370
inpatient hospitalization | 0.51 (0.87) | 0.43 (0.76) | 0.44 (0.79) | 0.40 (0.77) | 0.52 (0.81)
Statistical Analysis 1: Comparison: Nintedanib- Highly Adherent vs Nintedanib- Medium Adherent vs Nintedanib- Gradual Decliners vs Nintedanib- Intermediate Decliners vs Nintedanib- Rapid Decliners; [analysis description as in outcome 6, analysis 1]; Test type: Other; p = 0.270, ANOVA

28. Secondary Outcome: Beneficiary Characteristics -Inpatient Hospitalization Use and Spending: Inpatient Hosp - LOS According to Adherence Trajectories for the Idiopathic Pulmonary Fibrosis (IPF) Patients Who Were Initiated on Nintedanib
Description: The count of the number of days (length of stay (LOS)) a beneficiary was hospitalized in an inpatient facility during the baseline period, according to adherence trajectories for the idiopathic pulmonary fibrosis (IPF) patients who were initiated on nintedanib is reported.
  Length of stay for each inpatient hospitalization claim was calculated as the arithmetic difference between each claim's from and through dates.
Time Frame: as for outcome 2
Population: Eligible Patients set: All patients who met the criteria were included in the analysis dataset.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Nintedanib- Highly Adherent | Nintedanib- Medium Adherent | Nintedanib- Gradual Decliners | Nintedanib- Intermediate Decliners | Nintedanib- Rapid Decliners
Number analyzed (Participants) | 781 | 202 | 190 | 255 | 370
Days | 2.55 (5.82) | 2.03 (4.55) | 1.96 (3.97) | 1.99 (4.98) | 2.59 (5.24)
Statistical Analysis 1: Comparison: Nintedanib- Highly Adherent vs Nintedanib- Medium Adherent vs Nintedanib- Gradual Decliners vs Nintedanib- Intermediate Decliners vs Nintedanib- Rapid Decliners; [analysis description as in outcome 6, analysis 1]; Test type: Other; p = 0.306, ANOVA

29. Secondary Outcome: Beneficiary Characteristics - Inpatient Hospitalization Use and Spending: Inpatient Hosp. Spending - Total According to Adherence Trajectories for the Idiopathic Pulmonary Fibrosis (IPF) Patients Who Were Initiated on Nintedanib
Description: The total amount paid by all parties for all inpatient hospitalizations (for any cause) as reported in inpatient facility claims during the baseline period, according to adherence trajectories for the idiopathic pulmonary fibrosis (IPF) patients who were initiated on nintedanib is reported.
  This was calculated as the sum of the Medicare payment amount, the Medicare per diem amount, the non-Medicare payer amount, and the patient OOP amount.
Time Frame: as for outcome 2
Population: Eligible Patients set: All patients who met the criteria were included in the analysis dataset.
Measure: Mean (Standard Deviation); unit: United States Dollar
Arm/Group | Nintedanib- Highly Adherent | Nintedanib- Medium Adherent | Nintedanib- Gradual Decliners | Nintedanib- Intermediate Decliners | Nintedanib- Rapid Decliners
Number analyzed (Participants) | 781 | 202 | 190 | 255 | 370
United States Dollar | 6,721 (13,657) | 5,519 (12,920) | 5,011 (9,940) | 4,783 (10,904) | 6,323 (11,317)
Statistical Analysis 1: Comparison: Nintedanib- Highly Adherent vs Nintedanib- Medium Adherent vs Nintedanib- Gradual Decliners vs Nintedanib- Intermediate Decliners vs Nintedanib- Rapid Decliners; [analysis description as in outcome 6, analysis 1]; Test type: Other; p = 0.145, ANOVA

30. Secondary Outcome: Beneficiary Characteristics - Inpatient Hospitalization Use and Spending: Inpatient Hosp. Spending - OOP According to Adherence Trajectories for the Idiopathic Pulmonary Fibrosis (IPF) Patients Who Were Initiated on Nintedanib
Description: The total amount paid out-of-pocket (Inpatient hosp. spending - OOP) by the beneficiary for all inpatient hospitalizations (for any cause) as reported in inpatient facility claims during the baseline period, according to adherence trajectories for the idiopathic pulmonary fibrosis (IPF) patients who were initiated on nintedanib is reported.
Time Frame: as for outcome 2
Population: Eligible Patients set: All patients who met the criteria were included in the analysis dataset.
Measure: Mean (Standard Deviation); unit: United States Dollar
Arm/Group | Nintedanib- Highly Adherent | Nintedanib- Medium Adherent | Nintedanib- Gradual Decliners | Nintedanib- Intermediate Decliners | Nintedanib- Rapid Decliners
Number analyzed (Participants) | 781 | 202 | 190 | 255 | 370
United States Dollar | 555 (852) | 462 (750) | 485 (780) | 454 (832) | 604 (876)
Statistical Analysis 1: Comparison: Nintedanib- Highly Adherent vs Nintedanib- Medium Adherent vs Nintedanib- Gradual Decliners vs Nintedanib- Intermediate Decliners vs Nintedanib- Rapid Decliners; [analysis description as in outcome 6, analysis 1]; Test type: Other; p = 0.109, ANOVA

31. Secondary Outcome: Beneficiary Characteristics - Outpatient Facility Use and Spending: Outpatient Facility - Count According to Adherence Trajectories for the Idiopathic Pulmonary Fibrosis (IPF) Patients Who Were Initiated on Nintedanib
Description: The count of the number of unique dates with an outpatient facility (Outpatient facility - count) for any cause claim a beneficiary had during the baseline period, according to adherence trajectories for the idiopathic pulmonary fibrosis (IPF) patients who were initiated on nintedanib is reported.
Time Frame: as for outcome 2
Population: Eligible Patients set: All patients who met the criteria were included in the analysis dataset.
Measure: Mean (Standard Deviation); unit: Unique outpatient visit
Arm/Group | Nintedanib- Highly Adherent | Nintedanib- Medium Adherent | Nintedanib- Gradual Decliners | Nintedanib- Intermediate Decliners | Nintedanib- Rapid Decliners
Number analyzed (Participants) | 781 | 202 | 190 | 255 | 370
Unique outpatient visit | 8.25 (7.08) | 8.87 (8.59) | 8.35 (6.88) | 8.53 (8.27) | 9.13 (8.68)
Statistical Analysis 1: Comparison: Nintedanib- Highly Adherent vs Nintedanib- Medium Adherent vs Nintedanib- Gradual Decliners vs Nintedanib- Intermediate Decliners vs Nintedanib- Rapid Decliners; [analysis description as in outcome 6, analysis 1]; Test type: Other; p = 0.454, ANOVA

32. Secondary Outcome: Beneficiary Characteristics: Outpatient Facility Use and Spending: Outpatient Facility Spending - Total According to Adherence Trajectories for the Idiopathic Pulmonary Fibrosis (IPF) Patients Who Were Initiated on Nintedanib
Description: The total amount paid by all parties for outpatient facility claims during the baseline period, according to adherence trajectories for the idiopathic pulmonary fibrosis (IPF) patients who were initiated on nintedanib is reported. This was calculated as the sum of the Medicare payment amount, the blood deductible liability amount, the non-Medicare payer amount, and the patient OOP amount.
Time Frame: as for outcome 2
Population: Eligible Patients set: All patients who met the criteria were included in the analysis dataset.
Measure: Mean (Standard Deviation); unit: United States Dollar
Arm/Group | Nintedanib- Highly Adherent | Nintedanib- Medium Adherent | Nintedanib- Gradual Decliners | Nintedanib- Intermediate Decliners | Nintedanib- Rapid Decliners
Number analyzed (Participants) | 781 | 202 | 190 | 255 | 370
United States Dollar | 3,497 (10,264) | 3,623 (4,775) | 3,396 (4,684) | 3,711 (6,679) | 3,846 (6,756)
Statistical Analysis 1: Comparison: Nintedanib- Highly Adherent vs Nintedanib- Medium Adherent vs Nintedanib- Gradual Decliners vs Nintedanib- Intermediate Decliners vs Nintedanib- Rapid Decliners; [analysis description as in outcome 6, analysis 1]; Test type: Other; p = 0.960, ANOVA

33. Secondary Outcome: Beneficiary Characteristics - Outpatient Facility Use and Spending: Outpatient Facility Spending - OOP According to Adherence Trajectories for the Idiopathic Pulmonary Fibrosis (IPF) Patients Who Were Initiated on Nintedanib
Description: The total amount paid out-of-pocket by the beneficiary for services as reported in outpatient facility claims during the baseline period, according to adherence trajectories for the idiopathic pulmonary fibrosis (IPF) patients who were initiated on nintedanib is reported.
Time Frame: as for outcome 2
Population: Eligible Patients set: All patients who met the criteria were included in the analysis dataset.
Measure: Mean (Standard Deviation); unit: United States Dollar
Arm/Group | Nintedanib- Highly Adherent | Nintedanib- Medium Adherent | Nintedanib- Gradual Decliners | Nintedanib- Intermediate Decliners | Nintedanib- Rapid Decliners
Number analyzed (Participants) | 781 | 202 | 190 | 255 | 370
United States Dollar | 687 (1,095) | 742 (927) | 685 (810) | 762 (1,393) | 858 (1,666)
Statistical Analysis 1: Comparison: Nintedanib- Highly Adherent vs Nintedanib- Medium Adherent vs Nintedanib- Gradual Decliners vs Nintedanib- Intermediate Decliners vs Nintedanib- Rapid Decliners; [analysis description as in outcome 6, analysis 1]; Test type: Other; p = 0.265, ANOVA

34. Secondary Outcome: Beneficiary Characteristics -Home Health Use and Spending: Home Health - Count According to Adherence Trajectories for the Idiopathic Pulmonary Fibrosis (IPF) Patients Who Were Initiated on Nintedanib
Description: The count of the number of home health visits a beneficiary had during the baseline period, according to adherence trajectories for the idiopathic pulmonary fibrosis (IPF) patients who were initiated on nintedanib is reported. It was calculated by summing the total visit count on each claim across claims.
Time Frame: as for outcome 2
Population: Eligible Patients set: All patients who met the criteria were included in the analysis dataset.
Measure: Mean (Standard Deviation); unit: Home health visits
Arm/Group | Nintedanib- Highly Adherent | Nintedanib- Medium Adherent | Nintedanib- Gradual Decliners | Nintedanib- Intermediate Decliners | Nintedanib- Rapid Decliners
Number analyzed (Participants) | 781 | 202 | 190 | 255 | 370
Home health visits | 1.31 (5.88) | 0.90 (3.95) | 0.82 (3.78) | 1.38 (5.63) | 2.35 (9.31)
Statistical Analysis 1: Comparison: Nintedanib- Highly Adherent vs Nintedanib- Medium Adherent vs Nintedanib- Gradual Decliners vs Nintedanib- Intermediate Decliners vs Nintedanib- Rapid Decliners; [analysis description as in outcome 6, analysis 1]; Test type: Other; p = 0.026, ANOVA

35. Secondary Outcome: Beneficiary Characteristics - Home Health Use and Spending: Home Health Spending - Total According to Adherence Trajectories for the Idiopathic Pulmonary Fibrosis (IPF) Patients Who Were Initiated on Nintedanib
Description: The total amount paid by all parties (Home health spending - total) for home health claims during the baseline period, according to adherence trajectories for the idiopathic pulmonary fibrosis (IPF) patients who were initiated on nintedanib is reported.
  This was calculated as the sum of the Medicare payment amount, the blood deductible liability amount, the non-Medicare payer amount, and the patient OOP amount.
Time Frame: as for outcome 2
Population: Eligible Patients set: All patients who met the criteria were included in the analysis dataset.
Measure: Mean (Standard Deviation); unit: United States Dollar
Arm/Group | Nintedanib- Highly Adherent | Nintedanib- Medium Adherent | Nintedanib- Gradual Decliners | Nintedanib- Intermediate Decliners | Nintedanib- Rapid Decliners
Number analyzed (Participants) | 781 | 202 | 190 | 255 | 370
United States Dollar | 280 (1,080) | 232 (880) | 177 (738) | 286 (1,091) | 495 (1,797)
Statistical Analysis 1: Comparison: Nintedanib- Highly Adherent vs Nintedanib- Medium Adherent vs Nintedanib- Gradual Decliners vs Nintedanib- Intermediate Decliners vs Nintedanib- Rapid Decliners; [analysis description as in outcome 6, analysis 1]; Test type: Other; p = 0.016, ANOVA

36. Secondary Outcome: Beneficiary Characteristics - Part B Spending: Total According to Adherence Trajectories for the Idiopathic Pulmonary Fibrosis (IPF) Patients Who Were Initiated on Nintedanib
Description: The total amount paid by all parties for Carrier and Durable Medical Equipment claims during the baseline period, according to adherence trajectories for the idiopathic pulmonary fibrosis (IPF) patients who were initiated on nintedanib is reported. It was calculated as the sum of the allowed amounts on each claim.
Time Frame: as for outcome 2
Population: Eligible Patients set: All patients who met the criteria were included in the analysis dataset.
Measure: Mean (Standard Deviation); unit: United States Dollar
Arm/Group | Nintedanib- Highly Adherent | Nintedanib- Medium Adherent | Nintedanib- Gradual Decliners | Nintedanib- Intermediate Decliners | Nintedanib- Rapid Decliners
Number analyzed (Participants) | 781 | 202 | 190 | 255 | 370
United States Dollar | 7,136 (9,877) | 6,907 (7,229) | 7,446 (7,890) | 6,876 (4,857) | 6,916 (6,364)
Statistical Analysis 1: Comparison: Nintedanib- Highly Adherent vs Nintedanib- Medium Adherent vs Nintedanib- Gradual Decliners vs Nintedanib- Intermediate Decliners vs Nintedanib- Rapid Decliners; [analysis description as in outcome 6, analysis 1]; Test type: Other; p = 0.937, ANOVA

37. Secondary Outcome: Beneficiary Characteristics -Part B Spending: Part B Spending - OOP: According to Adherence Trajectories for the Idiopathic Pulmonary Fibrosis (IPF) Patients Who Were Initiated on Nintedanib
Description: The total amount paid out-of-pocket (Part B spending - OOP) by the beneficiary for Carrier and Durable Medical Equipment claims during the baseline period, according to adherence trajectories for the idiopathic pulmonary fibrosis (IPF) patients who were initiated on nintedanib is reported.
Time Frame: as for outcome 2
Population: Eligible Patients set: All patients who met the criteria were included in the analysis dataset.
Measure: Mean (Standard Deviation); unit: United States Dollar
Arm/Group | Nintedanib- Highly Adherent | Nintedanib- Medium Adherent | Nintedanib- Gradual Decliners | Nintedanib- Intermediate Decliners | Nintedanib- Rapid Decliners
Number analyzed (Participants) | 781 | 202 | 190 | 255 | 370
United States Dollar | 1,481 (1,962) | 1,432 (1,429) | 1,532 (1,484) | 1,428 (950) | 1,438 (1,259)
Statistical Analysis 1: Comparison: Nintedanib- Highly Adherent vs Nintedanib- Medium Adherent vs Nintedanib- Gradual Decliners vs Nintedanib- Intermediate Decliners vs Nintedanib- Rapid Decliners; [analysis description as in outcome 6, analysis 1]; Test type: Other; p = 0.948, ANOVA

38. Secondary Outcome: Beneficiary Characteristics - Total Spending: Total Medical Spending According to Adherence Trajectories for the Idiopathic Pulmonary Fibrosis (IPF) Patients Who Were Initiated on Nintedanib
Description: The total amount paid by all parties for all medical services during the baseline period, including inpatient, outpatient, home health and Part B, according to adherence trajectories for the idiopathic pulmonary fibrosis (IPF) patients who were initiated on nintedanib is reported.
Time Frame: as for outcome 2
Population: Eligible Patients set: All patients who met the criteria were included in the analysis dataset.
Measure: Mean (Standard Deviation); unit: United States Dollar
Arm/Group | Nintedanib- Highly Adherent | Nintedanib- Medium Adherent | Nintedanib- Gradual Decliners | Nintedanib- Intermediate Decliners | Nintedanib- Rapid Decliners
Number analyzed (Participants) | 781 | 202 | 190 | 255 | 370
United States Dollar | 17,634 (23,297) | 16,280 (18,712) | 16,029 (15,873) | 15,656 (16,455) | 17,581 (17,982)
Statistical Analysis 1: Comparison: Nintedanib- Highly Adherent vs Nintedanib- Medium Adherent vs Nintedanib- Gradual Decliners vs Nintedanib- Intermediate Decliners vs Nintedanib- Rapid Decliners; [analysis description as in outcome 6, analysis 1]; Test type: Other; p = 0.574, ANOVA

39. Secondary Outcome: Beneficiary Characteristics - Total Spending: All Spending - Total According to Adherence Trajectories for the Idiopathic Pulmonary Fibrosis (IPF) Patients Who Were Initiated on Nintedanib
Description: The total amount paid by all parties for all medical and pharmacy claims during the baseline period, according to adherence trajectories for the idiopathic pulmonary fibrosis (IPF) patients who were initiated on nintedanib is reported. Was calculated as the sum of total pharmacy and total medical spending.
Time Frame: as for outcome 2
Population: Eligible Patients set: All patients who met the criteria were included in the analysis dataset.
Measure: Mean (Standard Deviation); unit: United States Dollar
Arm/Group | Nintedanib- Highly Adherent | Nintedanib- Medium Adherent | Nintedanib- Gradual Decliners | Nintedanib- Intermediate Decliners | Nintedanib- Rapid Decliners
Number analyzed (Participants) | 781 | 202 | 190 | 255 | 370
United States Dollar | 21,304 (27,331) | 19,323 (19,660) | 18,928 (17,396) | 19,366 (18,723) | 21,377 (21,324)
Statistical Analysis 1: Comparison: Nintedanib- Highly Adherent vs Nintedanib- Medium Adherent vs Nintedanib- Gradual Decliners vs Nintedanib- Intermediate Decliners vs Nintedanib- Rapid Decliners; [analysis description as in outcome 6, analysis 1]; Test type: Other; p = 0.491, ANOVA

40. Secondary Outcome: Beneficiary Characteristics - Total Spending: All Spending - OOP According to Adherence Trajectories for the Idiopathic Pulmonary Fibrosis (IPF) Patients Who Were Initiated on Nintedanib
Description: The total amount paid out-of-pocket (OOP) by the beneficiary during the baseline period, according to adherence trajectories for the idiopathic pulmonary fibrosis (IPF) patients who were initiated on nintedanib is reported.
Time Frame: as for outcome 2
Population: Eligible Patients set: All patients who met the criteria were included in the analysis dataset.
Measure: Mean (Standard Deviation); unit: United States Dollar
Arm/Group | Nintedanib- Highly Adherent | Nintedanib- Medium Adherent | Nintedanib- Gradual Decliners | Nintedanib- Intermediate Decliners | Nintedanib- Rapid Decliners
Number analyzed (Participants) | 781 | 202 | 190 | 255 | 370
United States Dollar | 3,522 (3,209) | 3,367 (2,355) | 3,461 (2,555) | 3,452 (2,566) | 3,791 (3,027)
Statistical Analysis 1: Comparison: Nintedanib- Highly Adherent vs Nintedanib- Medium Adherent vs Nintedanib- Gradual Decliners vs Nintedanib- Intermediate Decliners vs Nintedanib- Rapid Decliners; [analysis description as in outcome 6, analysis 1]; Test type: Other; p = 0.432, ANOVA

ADVERSE EVENTS:
Time Frame: Adverse events were not collected.
Description: Given the information available within the Medicare claims database for this study, extraction on adverse events data was not conducted and only data related to the study objectives was extracted. Therefore, information about individual adverse events was not available. Only data on aggregate-level medication use were analyzed.
Arm/Group | Nintedanib
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
The use of administrative claims data restricted the ability to observe medication use, the only signal of use was from prescription drug claims, which do not provide any details of use and require the assumption that patients were adherent while they had medication supply. The follow-up period was limited to the first year after nintedanib initiation, therefore may not apply to adherence patterns after this period.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-12): https://cdn.clinicaltrials.gov/large-docs/84/NCT05022784/Prot_SAP_000.pdf